CLINICAL TRIAL: NCT01237210
Title: Magnetic Resonance Spectroscopy of Parkinson's Disease at 7 Tesla
Brief Title: 7T MRS in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0803M28421
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; PD; magnetic resonance spectroscopy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is looking for healthy controls and patients with Parkinson's (PD) to perform an MR scan.

1. The neurochemical profile of the SN of patients with PD as measured by high field MRS will differ from that of healthy controls, in that glutathione will be lower due to oxidative stress, lactate will be higher due to mitochondrial dysfunction, the gliosis markers myo-inositol and glutamine will be higher due to inflammation (glial activation) and N-acetylaspartate and glutamate will be lower due to neuronal loss/damage.
2. There will be a relationship between neurochemical changes and disease severity.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's disease Group

* Parkinson's disease (clinical diagnostic criteria)
* Age 45-75 years inclusive
* Able to safely undergo MRI scanning
* Absence of diabetes and smoking
* Capable of giving informed consent

Healthy Control Group

* Age 45-75 years inclusive
* Able to safely undergo MRI scanning
* Absence of diabetes and smoking
* Capable of giving informed consent

Exclusion Criteria:

Parkinson's disease Group

* Dementia (clinically determined by PI Dr. Tuite)
* Diagnosis of atypical parkinsonism
* Inability to safely undergo MRI scanning
* Inability to give informed consent
* Unstable medical conditions
* Present smoker
* Diabetic (on oral or injectable medications for diabetes)
* Taken coenzyme Q10 or Vitamin E in the 2 weeks prior to the scan
* Does not meet age criteria

Healthy Control Group

* Has a 1st degree relative with PD
* Dementia (clinically determined by PI Dr. Tuite)
* Inability to safely undergo MRI scanning
* Inability to give informed consent
* Unstable medical conditions
* Present smoker
* Diabetic (on oral or injectable medications for diabetes)
* Taken coenzyme Q10 or Vitamin E in the 2 weeks prior to the scan
* Does not meet age criteria

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance spectroscopy (MRS) | Baseline
  We will utilize optimized magnetic resonance spectroscopy (MRS) methodology to address theories of pathogenesis of Parkinson's disease (PD) by quantifying glutathione (GSH), lactate, glutamine and myo-inositol levels of the unilateral substantia nigra (SN) of healthy volunteers and patients with PD.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tuite, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota/CMRR, Minneapolis, Minnesota, United States